CLINICAL TRIAL: NCT04157699
Title: An Open-Label Phase 2 Study to Evaluate Safety and Efficacy of QL-007 Tablets in Combination With Tenofovir in Naive Patients With Chronic Hepatitis b: a Multicenter, Randomized, Positive Controlled Clinical Trial
Brief Title: An Study to Evaluate Safety and Efficacy of QL-007 Tablets in Combination With Tenofovir in Naive Patients With Chronic Hepatitis b
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL-007-201
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis b
Keywords: HBeAg-positive chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- QL-007 100 mg QD + TDF (Experimental): QL-007 tablet 100 mg QD was combined with TDF tablet 300mg
  Interventions: Drug: TDF tablet; Drug: QL-007
- QL-007 200 mg QD + TDF (Experimental): QL-007 tablets 200 mg QD were combined with TDF tablet 300mg
  Interventions: Drug: TDF tablet; Drug: QL-007
- QL-007 400 mg QD+ TDF (Experimental): QL-007 tablets 400 mg QD were combined with TDF tablet 300mg
  Interventions: Drug: TDF tablet; Drug: QL-007
- QL-007 200 mg BID+ TDF (Experimental): QL007 tablets 200 mg BID were combined with TDF tablet 300mg
  Interventions: Drug: TDF tablet; Drug: QL-007
- TDF monotherapy (Active Comparator): TDF tablet 300mg
  Interventions: Drug: TDF tablet

INTERVENTIONS:
Drug: TDF tablet — TDF tablet 300mg QD
  Other Names: Tenofovir disoproxil fumarate tablet
Drug: QL-007 — QL-007 tablet
  Arms: QL-007 100 mg QD + TDF; QL-007 200 mg BID+ TDF; QL-007 200 mg QD + TDF; QL-007 400 mg QD+ TDF

SUMMARY:
This is an open label, randomized, multi-center, comparative study. Subjects will be screened prior to study entry to establish eligibility. 100 Subjects who meet all the selection criteria will be randomly assigned 1:1:1:1:1 to (A) QL007 100 mg QD+ Tenofovir dipirofurate fumarate （TDF）300 mg QD, (B) QL007 200 mg QD+ TDF 300 mg QD, (C) QL007 400 mg QD+ TDF 300 mg QD, (D) QL007 200 mg BID+ TDF 300 mg QD, (E) TDF 300 mg QD.

The purpose of this study was to evaluate the efficacy and safety of QL-007 in combination with TDF in HBeAg positive patients with chronic hepatitis b, and to recommend a reasonable regimen for phase III study.

DETAILED DESCRIPTION:
The subjects received the drug treatment for a total of 96 weeks, which was divided into two stages: the first stage: 0-24 weeks as the core treatment period and 25-48 weeks as the extended treatment period. The second stage: 49-96 weeks is the extended treatment period，subjects will enter the second stage of treatment according to the dose of the first stage. When the efficacy data of the first phase determine the optimal dose of QL-007, all subjects entering the second phase will receive the optimal dose of QL-007 and continue treatment with tenofovir dipirofurate fumarate (QL-007 XX mg+TDF) for the second phase 49-96 weeks of extended treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years (inclusive) with chronic HBV infection prior to baseline;
2. Positive for HBeAg;
3. Patients who had not previously received anti-HBV treatment (including nucleoside or interferon) or had not received antiviral treatment for HBV (including nucleoside or interferon) within 6 months prior to the first taking the study drug;
4. HBV DNA≥20,000 IU/mL;
5. ALT levels > upper limit of normal value (ULN) and<5 times ULN;
6. Participants must have understood and signed the ICF.

Exclusion Criteria:

1. Known co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis D virus (HDV);
2. History of liver disease other than chronic hepatitis B, which may affect the judgment of the effectiveness or safety of the study drug
3. History of Gilbert's Disease;
4. History of decompensated liver disease or any sign of decompensated liver disease in the screening period;
5. Evidence of moderate or severe fibrosis or cirrhosis;
6. Evidence of HCC or AFP > 50 ng / ml in the screening period ;
7. Any Clinical laboratory values meet certain standards in the screening period;
8. subjects have clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months);
9. Risks of serious kidney and respiratory diseases;
10. Impaired gastrointestinal (GI) function or GI disease that may alter absorption of QL-007 as determined by the Investigator;
11. Receiving medications that meet one of the following criteria and that cannot be discontinued ≥1 week prior to the start of treatment QL-007:

    * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes;
    * Moderate or strong inhibitors or strong inducers of CYP3A4
12. Intake of any drugs that can reduce enzyme activity;
13. History of bleeding diathesis;
14. Risks of mental and nervous system diseases during screening;
15. Pregnant or lactating female subjects; Female subjects of childbearing age who were not willing to use effective contraception throughout the study period or male subjects whose partners were fertile but were not willing to use effective contraception;
16. Volunteers who took an Investigational Product within 3 months or who have been within 5 half-lives of other trial drugs before the randomization.
17. Any other condition , which in the opinion of investigator would make a patient unfit for participation in a clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of QL-007 in combination with TDF in patients with HBeAg-positive chronic hepatitis b: HBV DNA level | 24 weeks
  The change of HBV DNA level at week 24 of treatment compared to baseline

SECONDARY OUTCOMES:
serological indexs | 96 weeks
  The changes of HBsAg and HBeAg level from baseline at week 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96
serological indexs | 96 weeks
  The percentage of subjects with HBsAg and HBeAg serological clearance and/or seroconversion at week 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96
Virological indexs | 96 weeks
  The changes of HBV DNA level compared to baseline at week 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96
Virological indexs | 96 weeks
  The rate of HBV DNA negative subjects (HBV DNA <60 IU/mL) at week 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96
biochemistry index | 96 weeks
  The changes of ALT at week 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96 compared to baseline
biochemistry index | 96 weeks
  The percentage of subjects with normal ALT level at weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84 and 96
Other evaluation indexes of pharmacodynamics exploration | 96 weeks
  The changes of HBV RNA and HBcrAg level compared with baseline at week 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84 and 96
To evaluate the tolerance of QL-007 in combination with TDF: incidence of adverse events | 96 weeks
  The incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, PhD, Principal Investigator — Southern Hospital of Southern Medical University; Junqi Niu, PhD, Principal Investigator — The First Hospital of Jilin University
Locations (2):
- China (2):
  - Southern Hospital of Southern Medical University, Guangzhou, Guangdong
  - The first hospital of Jilin university, Changchun, Jilin